CLINICAL TRIAL: NCT05409079
Title: Schulze Muscular Dystrophy Ability Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AbiliTech Medical Inc. (Industry)
Collaborators: Richard M. Schulze Family Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Schulze
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Muscular Dystrophies; Spinal Muscular Atrophy; Duchenne Muscular Dystrophy; Limb Girdle Muscular Dystrophy; FSHD; Cerebral Palsy; Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophies; Muscular Atrophy, Spinal; Muscular Dystrophy, Duchenne; Muscular Dystrophies, Limb-Girdle; Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Abilitech Assist (Experimental): The Abilitech™ Assist device is a passively powered orthotic device designed to support and assist the arms of patients with neuromuscular weakness for activities of daily living.
  Interventions: Device: Abilitech Assist

INTERVENTIONS:
Device: Abilitech Assist — The Abilitech™ Assist is an externally worn device supported by a body frame, which is designed to support and assist the arms in activities of daily living (ADL's). The Abilitech Assist is comprised of three parts: a modular body vest that adjusts to accommodate different body sizes, a single arm orthosis that attaches to the body vest, and an external power pack and controller for tensioning the arm's internal springs to adjust the arm's level of assist. The device augments a user's native arm function to provide lift assistance. Software customizes the spring tension for the level of assist required. The user can turn the system ON/OFF and toggle and adjust the level of assist (e.g., low, medium or high assist) using a pushbutton controller.

SUMMARY:
The primary objective of the Schulze study is to evaluate the function of the upper limbs of subjects diagnosed with neuromuscular disorders, with and without use of the Abilitech Assist device in the clinic and home environments. Functional outcomes will include documenting active range of motion and the ability to perform activities of daily living (ADLs) using the standardized Canadian Occupational Performance Measure (COPM) and the Role Evaluation of Activities of Life (REAL) assessments. Secondary objectives are to assess the safety record and report on adverse events (AEs) and parameters related to device usage, including device usage time and the time required to don/doff the device. Secondary objectives also include characterization of user upper limb performance based on etiology.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between 10 and 99 years of age, with onset of neuromuscular conditions that cause quadriparesis
2. MMT score of 1-3 in the elbow, wrist and hand; and a MMT score of 2-3 in the shoulder of at least one of the subject's arms
3. Ability of subject to raise their forearm off of their lap or laptray
4. Willingness to comply and participate with the study protocol and attend the study sessions
5. Ability to communicate verbally and respond to questions and commands
6. Ability to provide informed consent
7. Selected for participation based on investigator discretion

Exclusion Criteria:

1. Use of invasive ventilator
2. Open wounds or chronic pressure sores on upper extremities, neck, back or torso
3. Significantly unstable upper extremity joints
4. Unhealed bone fractures in the upper extremities
5. Active rotator cuff tear, grade 2 or 3
6. Surgical fixations limiting full passive range of motion
7. Uncontrolled upper-limb spasticity that significantly limits normal range of motion
8. Uncontrollable pain in the neck, shoulders or upper limbs
9. Ability to fully raise both hands simultaneously above their head with ease as defined by the investigator
10. Lack passive shoulder abduction of 120 degrees
11. Lack 90 degrees of passive elbow extension
12. Unable to follow instructions
13. Exhibit significant behavioral problems
14. Inability to provide consent

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Change from Baseline before device intervention (30 days), and after device intervention (60 days)
  The Canadian Occupational Performance Measure is an evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time. The COPM results in two main scores - PERFORMANCE and SATISFACTION - each out of 10. PERFORMANCE and SATISFACTION scores can be generated for up to 5 individual occupational performance problems. Average PERFORMANCE and SATISFACTION scores can be calculated by summing individual problem scores and dividing by the number of problems. Change in scores for both PERFORMANCE and SATISFACTION can be calculated after a reassessment interval and a comparison of individual's score differences from Time 1 (assessment) to Time 2 (re-assessment). Increases in scores indicate improvement in task performance and satisfaction.
Roll Evaluation of Activities of Life (REAL) assessment | Change from Baseline before device intervention (30 days), and after device intervention (60 days)
  The REAL is an instrument to help professionals assess an individuals ability to care for themselves at home, at school and in the community. This assessment includes 136 total items with two domains(ADL: 78 items, IADL:58 items) that are rated using a 4-point scale (0-3) to describe whether an individual is unable, sleds, occasionally, or frequently able to complete a task. Scores are summed for each domain and compared over time with increases in scores indicating improvement in each domain.

CONTACTS AND LOCATIONS:
Locations (1):
- Gillette Children's, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided